CLINICAL TRIAL: NCT06171438
Title: Molecular Markers of Acute Kidney Injury in Elderly Deceased Donors
Acronym: MoliDon
Status: Completed | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of Department of Nephrology and Transplant Center, Institute for Clinical and Experimental Medicine
Other Study IDs: G339-2021
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Kidney Transplantation; Acute Kidney Injury
Keywords: kidney transplantation; donor kidney; microarray
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — donor and recipient kidney biopsies, urine and blood samples of donor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Acute kidney injury (AKI): Donors with AKI (acute kidney injury) defined based on the results of creatinine increase and diuresis decrease before organ harvest.
  Interventions: Diagnostic Test: Urine Biomarkers; Diagnostic Test: Gene expression profiling of donor kidneys by microarray; Diagnostic Test: Gene expression profiling of recipient kidneys by microarray
- no-AKI: Donors without AKI (acute kidney injury) defined based on the results of creatinine increase and diuresis decrease before organ harvest.
  Interventions: Diagnostic Test: Urine Biomarkers; Diagnostic Test: Gene expression profiling of donor kidneys by microarray; Diagnostic Test: Gene expression profiling of recipient kidneys by microarray
- delayed graft function (DGF): Donors and the paired recipients in whom the organ was transplanted in IKEM (Institute for Clinical and Experimental Medicine) who developed delayed graft function (DGF) defined as dialysis in the 1st week after transplantation.
  Interventions: Diagnostic Test: Urine Biomarkers; Diagnostic Test: Gene expression profiling of donor kidneys by microarray; Diagnostic Test: Gene expression profiling of recipient kidneys by microarray
- no-DGF: Donors and the paired recipients in whom the organ was transplanted in IKEM (Institute for Clinical and Experimental Medicine) with immediate graft function (no-DGF).
  Interventions: Diagnostic Test: Urine Biomarkers; Diagnostic Test: Gene expression profiling of donor kidneys by microarray; Diagnostic Test: Gene expression profiling of recipient kidneys by microarray
- Recipient IFTA: Donors and the paired recipients in whom the organ was transplanted in IKEM with 3-month protocol biopsy histology finding of IFTA≥2.
  Interventions: Diagnostic Test: Gene expression profiling of donor kidneys by microarray; Diagnostic Test: Gene expression profiling of recipient kidneys by microarray
- Recipient no-IFTA: Donors and the paired recipients in whom the was transplanted in IKEM with 3-month protocol biopsy histology finding of IFTA<2.
  Interventions: Diagnostic Test: Gene expression profiling of donor kidneys by microarray; Diagnostic Test: Gene expression profiling of recipient kidneys by microarray

INTERVENTIONS:
Diagnostic Test: Urine Biomarkers — Biomarkers of kidney damage in donors, such as neutrophil gelatinase-associated lipocalin (NGAL), N-acetyl-beta-D-glucosaminidase (NAG), beta2-microglobulin, alpha1-microglobulin, alpha2-macroglobulin and transferrin will be measured by ELISA.
  Groups: Acute kidney injury (AKI); delayed graft function (DGF); no-AKI; no-DGF
Diagnostic Test: Gene expression profiling of donor kidneys by microarray — Gene expression profiling of donor kidney biopsies using Affymetrix microarray platform (PrimeView Human Gene Expression Array).
Diagnostic Test: Gene expression profiling of recipient kidneys by microarray — Gene expression profiling of donor kidney biopsies using Affymetrix microarray platform (PrimeView Human Gene Expression Array).

SUMMARY:
Scoring systems that combine donor clinical and morphological parameters to predict outcome of kidney transplantation lack enough specificity to be generally accepted. Compare to classical histology, molecular assessment of renal tissue offers unbiased and technically robust approach. In this prospective 3-months' observational study procurement biopsies in 180 brain death donors will be performed. Using microarray which detect top differently regulated genes, conventional histology, urinary AKI biomarkers, renal function and clinical variables models predicting DGF and early graft scarring (IFTA, poor graft function) in recipients will be constructed. The associations of AKI in donors with distinct fibrosis atrophy and AKI molecular signals will be found. Molecular techniques and final models may help to improve the decision-making process for the acceptance of kidneys from marginal donors but more importantly, it may help clinicians to guide less toxic immunosuppression in identified problematic grafts.

DETAILED DESCRIPTION:
The aim is to create a prediction model of early clinical outcome (delayed graft function) based on donor and recipient clinical variables, donor eGFR, urinary AKI biomarkers, histology (glomerulosclerosis, interstitial fibrosis, vascular changes) and top differently regulated genes found in microarray of wedge procurement donor biopsy. Construct a model capable to predict early renal allograft scarring (IFTA>2), and impaired graft function (eGFR<45 mL/min), as early as at 3 months. Describe renal molecular changes associated with established AKI in brain-death deceased donor and with aging.

ELIGIBILITY:
Inclusion Criteria:

* All DBD (donation after brain death) donors whose kidneys will be procured by transplant team of Institute for Clinical and Experimental Medicine (IKEM) in donor hospital.
* All DBD (donation after brain death) donors whose kidneys will be procured by transplant team of Institute for Clinical and Experimental Medicine (IKEM) at IKEM.

Exclusion Criteria:

* Donors with circulatory death
* Donors with machine perfusion
* Donors with multiorgan transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All DBD donors whose kidneys will be procured by IKEM transplant team either in donor hospital or at IKEM. Corresponding recipients, transplanted at IKEM will be further monitored. Patients will receive standard immunosuppression based on tacrolimus, mycophenolate mofetil and steroids along with induction (basiliximab in low risk and rATG in high-risk) according to center protocol. All procedures in transplant recipients will be routine ones, included for cause biopsies and 3M protocol biopsy (standard of care in the center).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Kidney graft function at month 3 | 3 months
  Kidney graft function is measured as estimated glomerular filtration in ml/s/1.73m2.

SECONDARY OUTCOMES:
Kidney graft survival | 1 year
  Measured as numbers of patients with graft loss censored to death.
Delayed graft function | 1 week
  The need of dialysis in the 1st week after transplantation. Measured as numbers of patients.
Fibrosis grade at month 3 | 3 months
  Histologic result of interstitial fibrosis and atrophy at protocol biopsy. Min 0, Max 3, higher means worse
Gene expression in Donor kidney | 3 months
  Whole transcriptome microarray profiling of wedge biopsy taken immediately after organ procurement.
Gene expression in 3-month protocol biopsy of recipient | 3 months
  Whole transcriptome microarray profiling of 3-months protocol biopsies of recipients .
Urinary biomarkers of AKI in donors before organ taking | 3 months
  NGAL, Neutrophil gelatinase-associated lipocalin, ng/ml.
Urinary biomarkers of AKI in donors before organ taking (NAG) | 3 months
  NAG, N-acetyl-beta-D-glucosamine, in IU/l
Urinary biomarkers of AKI in donors before organ taking (beta 2 microglobulin) | 3 months
  beta 2 microglobulin, in mg/l
Urinary biomarkers of AKI in donors before organ taking (alfa1 microglobulin) | 3 months
  alfa1 microglobulin, in mg/l
Urinary biomarkers of AKI in donors before organ taking (alfa2 macroglobulin) | 3 months
  alfa2 macroglobulin, in mg/l
Urinary biomarkers of AKI in donors before organ taking (transferrin) | 3 months
  transferrin, in mg/l

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Viklicky, Prof., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia